CLINICAL TRIAL: NCT05463952
Title: A PHASE I, OPEN-LABEL STUDY TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF ARV-471 (PF-07850327), A SINGLE AGENT IN JAPANESE PARTICIPANTS WITH ER+/HER2-LOCALLY ADVANCED OR METASTATIC BREAST CANCER
Brief Title: A Study to Learn About the Vepdegestrant (ARV-471, PF-07850327) in People With ER+/HER2- Locally Advanced or Metastatic Breast Cancer (BC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4891016
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vepdegestrant (Experimental): Daily oral dosages of vepdegestrant
  Interventions: Drug: vepdegestrant

INTERVENTIONS:
Drug: vepdegestrant — ARV-471 will be administered orally QD with food, in continuous dosing over 28-day cycles.
  Other Names: ARV-471; PF-07850327

SUMMARY:
The purpose of this clinical trial is to learn about the safety, tolerability, Pharmacokinetics (PK), and preliminary efficacy of ARV-471 as monotherapy in Japanese participants with ER+/HER2- locally advanced or metastatic breast cancer (mBC).

ELIGIBILITY:
Inclusion Criteria:

1. Participants (women and men) at least 20 years of age at the time of signing the informed consent.
2. Histological or cytological diagnosis of ER+/HER2- advanced breast cancer that is metastatic, recurrent, or locally advanced unresectable breast cancer.
3. Participants who are resistant to standard therapy or for which no standard therapy is available or have received.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Infromed Consent Document (ICD) and in this protocol.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
6. Adequate Bone Marrow or Coagulation Function.
7. Adequate Renal Function, defined as an estimated creatinine clearance ≥60 mL/min as calculated using the method standard for the institution.
8. Adequate Liver Function.
9. Participants with brain metastases must meet all the specified conditions.
10. Resolution of acute effects of any prior therapy to either baseline severity or CTCAE version 5.0 Grade ≤1.

Exclusion Criteria:

1. Participants with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix, Bowen's disease.
2. Participants sustaining major surgery defined as a complex procedure performed under regional or general anesthesia with a recovery period of at least 4 weeks prior to study enrollment.
3. Known or suspected hypersensitivity or severe allergy to active ingredient/excipients of ARV-471.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow. Palliative radiation for the alleviation of pain due to bone metastasis will be allowed during the study.
6. Concurrent administration of medications, foods or herbal supplements that are strong inhibitors or inducers of CYP3A4 and drugs with a known risk of causing Torsade de Pointes or QT interval prolongation. Prior use of strong CYP3A inhibitors and drugs with a known risk of causing Torsade de Pointes or QT interval prolongation must be stopped 7 days before enrollment and strong CYP3A inducers must be stopped 14 days before enrollment.
7. Prior treatment with ARV-471.
8. Systemic anticancer therapy chemotherapy or endocrine therapy within 14 days prior to study entry (6 weeks for mitomycin C or nitrosoureas). If the last immediate anticancer treatment contained an antibody-based agent(s) (approved or investigational), then an interval of 28 days or 5 half-lives (whichever is shorter) of the agent(s) prior to receiving the study intervention treatment is required.
9. Participants who have initiated therapy with bone-modifying agents (bisphosphonates, denosumab, or similar) within 14 days of enrollment.
10. Previous high-dose chemotherapy requiring stem cell rescue.
11. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry. A participant may be eligible even if they are in the follow-up phase of an investigational study as long as they haven't received treatment in the study for 5 half lives of the agents.
12. Serum pregnancy test (for females of childbearing potential) positive at screening and/or a breastfeeding participant.
13. Participants with active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), and known Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)-related illness.
14. Baseline standard 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
15. Any of the following in the previous 12 months: myocardial infarction, long QT syndrome, Torsade de Pointes, clinically important atrial or ventricular arrhythmias, serious conduction system abnormalities, unstable angina, coronary/peripheral artery bypass graft, symptomatic CHF, New York Heart Association class III or IV, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, and/or other clinical significant episode of thrombo-embolic disease. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, atrial fibrillation of any grade . If a participant has a cardiac rhythm device/pacemaker placed and QTcF >470 ms, the participant may be considered eligible. Participants with cardiac rhythm device/pacemaker must be discussed in detail with the sponsor to judge eligibility.
16. History of symptomatic cardiac valve disease.
17. Active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease or previous gastric resection or lap band surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2025-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Iwata H, Naito Y, Hattori M, Yoshimura A, Yonemori K, Aizawa M, Mori Y, Yoshimitsu J, Umeyama Y, Mukohara T. Safety and pharmacokinetics of vepdegestrant in Japanese patients with ER+ advanced breast cancer: a phase 1 study. Int J Clin Oncol. 2025 Jan;30(1):72-82. doi: 10.1007/s10147-024-02648-3. Epub 2024 Nov 20. PMID 39565495
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese participants with estrogen receptor (ER+) or human epidermal growth factor receptor 2 (HER-2) locally advanced or metastatic breast cancer (mBC) were treated with ARV-471 (PF-07850327) as monotherapy. A total of 6 participants were enrolled.
Pre-assignment Details: Results are reported at primary completion date. Remaining results would be reported on completion of analysis at study completion date later.
Groups:
- ARV-471 200 mg: Participants received ARV-471 200 milligrams (mg) orally once daily (QD) with food, in continuous dosing over 28-day cycle (1 cycle = 28 days). Participants continued treatment at the discretion of the investigator until a treatment discontinuation criterion was met (disease progression; global deterioration of health status requiring discontinuation; unacceptable toxicity; pregnancy; significant protocol violation; lost to follow-up; participant refused further treatment; study terminated by sponsor; death).
Period: Treatment
Arm/Group | ARV-471 200 mg
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive disease | 4
Not completed — Ongoing | 2
Period: Follow-up
Arm/Group | ARV-471 200 mg
Started | 4 (Participant who discontinued treatment but were followed-up for safety.)
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who have been assigned to ARV-471.
Groups:
- ARV-471 200 mg: Participants received ARV-471 200 mg orally QD, in continuous dosing over 28-day cycle.
Arm/Group | ARV-471 200 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (6.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLTs) During First Treatment Cycle
Description: DLT was defined as any adverse event (AE) or abnormal laboratory value which were related to ARV-471 and assessed as unrelated to disease, disease progression, intercurrent illness or concomitant medications/therapies occurring during the first 28 days of treatment that met at least 1 of the study specified criteria.
Time Frame: Cycle 1 (28 days)
Population: DLT evaluable analysis set included all enrolled participants who received at least 75% of the planned dose intensity of study treatment and either experienced DLT or did not have major protocol deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | ARV-471 200 mg
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Participants With AEs and Serious AEs (SAEs)- All Causalities and Treatment Related
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness was judged by investigator. SAE was an AE resulted in any of the following outcomes: death, inpatient hospitalization or prolongation of existing hospitalization; was life-threatening experience (immediate risk of dying); resulted in persistent or significant disability/incapacity; congenital anomaly, a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic.
Time Frame: Day 1 of study treatment up to 35 days after last dose of study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

3. Secondary Outcome: Number of Participants With Laboratory Hematology Results by Maximum National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade
Description: The following hematology parameters were assessed: hemoglobin, platelets, white blood cell (WBC), absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils and absolute basophils. Laboratory abnormality events were graded according to NCI CTCAE v 5.0 (grade 0=no change from normal or reference range, grade 1=mild, grade 2= moderate, grade 3= severe, grade 4= life-threatening and grade 5= death related).
Time Frame: During study treatment, approximately 1.5 years
Reporting Status: Not Posted, anticipated posting 2024-09

4. Secondary Outcome: Number of Participants With Laboratory Chemistry Results by Maximum NCI-CTCAE Grade
Description: The following chemistry parameters were assessed: aspartate transaminase (AST), alkaline phosphatase (ALP), sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen (BUN) or urea, creatinine, uric acid, glucose (non-fasted), albumin, phosphorus or phosphate, creatinine kinase (CK), amylase and lipase. Laboratory abnormality events were graded according to NCI CTCAE v 5.0 (grade 0=no change from normal or reference range, grade 1=mild, grade 2= moderate, grade 3= severe, grade 4= life-threatening and grade 5= death related).
Time Frame: During study treatment, approximately 1.5 years
Reporting Status: Not Posted, anticipated posting 2024-09

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time Tau (AUCtau) of ARV 471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

8. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

9. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

10. Secondary Outcome: Metabolite Ratio for Cmax (MRCmax)
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

11. Secondary Outcome: Metabolite Ratio for AUCtau (MRAUCtau)
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

12. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

13. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

14. Secondary Outcome: Apparent Total Clearance (CL/F) of ARV-471
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of ARV-471
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

16. Secondary Outcome: Effective Half-Life Based on Accumulation Ratio (t½Eff) of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

17. Secondary Outcome: Accumulation Ratio (Rac) Based on AUC of ARV-471 and ARV-473
Time Frame: Through the end of the study treatment (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

18. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) and partial response (PR) as per Response Evaluation Criteria in Solid Tumours (RECIST version [v] 1.1). BOR: best response was recorded from start of study treatment until disease progression or death due to any cause. CR: complete disappearance of all target lesions with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<]10 millimeter [mm]). PR: greater than or equal to (>=) 30 percent (%) decrease under baseline of sum of diameters of all targets measurable lesions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions. All target lesions were assessed.
Time Frame: From start of study treatment until disease progression or death due to any cause (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

19. Secondary Outcome: Clinical Benefit Response (CBR)
Description: CBR is defined as the percentage of participants with BOR of CR, PR and stable disease (SD) of 24 weeks duration or longer. As per RECIST v1.1. SD: Does not qualify for CR, PR or Progression. All target lesions must be assessed. Stable could follow PR only in the rare case that the sum increased by <20% from the nadir, but enough that a previously documented 30% decrease no longer held. CR: complete disappearance of all target lesions and non-target disease, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal short axis <10 mm). No new lesions. PR: >= 30% decrease under baseline of sum of diameters of all targets measurable lesions. Short diameter was used in sum for target nodes, while longest diameter was used in sum for all other target lesions.
Time Frame: From start of study treatment until disease progression or death due to any cause (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

20. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment (ie, start date) to the date of progression of disease (PD) or death due to any cause, whichever occurred first. PFS data was censored on the date of the last adequate tumor assessment for participants without an event (PD or death), for participants who started new anti-cancer treatment prior to an event, or for participants with an event after two or more missing tumor assessments. PD as per RECIST v1.1 for target lesions was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm. For non-target lesions- PD was defined as unequivocal progression of pre-existing lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until disease progression or death due to any cause or censoring date (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

21. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first in participants with confirmed objective response (CR or PR). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause (approximately 1.5 years)
Reporting Status: Not Posted, anticipated posting 2024-09

ADVERSE EVENTS:
Time Frame: Day 1 of study treatment up to 35 days last dose of study treatment (maximum up to 33 weeks as maximum treatment exposure was 28 weeks)
Arm/Group | ARV-471 200 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARV-471 200 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT05463952/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT05463952/SAP_001.pdf